CLINICAL TRIAL: NCT01114542
Title: A Trial Evaluating the Pharmacodynamic Response of NN1250 at Steady State Conditions in Subjects With Type 1 Diabetes
Brief Title: A Trial Evaluating the Effect of NN1250 at Steady State Conditions in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-1993; 2009-015897-36 (EudraCT Number); U1111-1113-6772 (Other: WHO)
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- IDeg 0.4 U/kg (Experimental)
  Interventions: Drug: insulin degludec
- IDeg 0.6 U/kg (Experimental)
  Interventions: Drug: insulin degludec
- IDeg 0.8 U/kg (Experimental)
  Interventions: Drug: insulin degludec
- IGlar 0.4 U/kg (Active Comparator)
  Interventions: Drug: insulin glargine
- IGlar 0.6 U/kg (Active Comparator)
  Interventions: Drug: insulin glargine
- IGlar 0.8 U/kg (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Subjects were randomised to one of three possible dose levels (low, middle or high) and to one of two treatment sequences. A treatment sequence consisted of 2 periods of each 13 days. One dose once daily. The trial products were administered subcutaneously (under the skin)
  Arms: IDeg 0.4 U/kg; IDeg 0.6 U/kg; IDeg 0.8 U/kg
Drug: insulin glargine — Subjects were randomised to one of three possible dose levels (low, middle or high) and to one of two treatment sequences. A treatment sequence consisted of 2 periods of each 13 days. One dose once daily. The trial products were administered subcutaneously (under the skin)
  Arms: IGlar 0.4 U/kg; IGlar 0.6 U/kg; IGlar 0.8 U/kg

SUMMARY:
This trial was conducted in Europe. The aim of this clinical trial was to evaluate the effect on the blood glucose-lowering effect of NN1250 (insulin degludec) in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Current total daily insulin treatment lower than 1.2 (I)U/kg/day
* Body mass index 18.0-28.0 kg/m^2

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period
* Supine blood pressure at screening (after resting for 5 min) outside the range of 90-140 mmHg for systolic or 50-90 mmHg for diastolic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-05-03 (Actual); Primary Completion 2010-08-10 (Actual); Study Completion 2010-08-10 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve during one dosing interval of Insulin Degludec at steady state | 0-24 hours after dosing on day 8

SECONDARY OUTCOMES:
Area under the glucose infusion rate curve during one dosing interval of insulin glargine at steady state | 0-24 hours after dosing on day 8
Area under the concentration-time curve during one dosing interval at steady state for Insulin Degludec | 0-24 hours after dosing on day 8
Area under the concentration-time curve during one dosing interval at steady state for insulin glargine | 0-24 hours after dosing on day 8

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Korsatko S, Nosek L, Coester HV, Deller S, Roepstorff C, Segel S, Kapur R, Haahr H, Hompesch M. Steady state is reached within 2-3 days of once-daily administration of degludec, a basal insulin with an ultralong duration of action. J Diabetes. 2016 Jan;8(1):132-8. doi: 10.1111/1753-0407.12266. Epub 2015 Mar 24. PMID 25581159
- [Result] Heise T, Hovelmann U, Nosek L, Hermanski L, Bottcher SG, Haahr H. Comparison of the pharmacokinetic and pharmacodynamic profiles of insulin degludec and insulin glargine. Expert Opin Drug Metab Toxicol. 2015;11(8):1193-201. doi: 10.1517/17425255.2015.1058779. Epub 2015 Jun 18. PMID 26086190
- [Result] Heise T, Kaplan K, Haahr HL. Day-to-Day and Within-Day Variability in Glucose-Lowering Effect Between Insulin Degludec and Insulin Glargine (100 U/mL and 300 U/mL): A Comparison Across Studies. J Diabetes Sci Technol. 2018 Mar;12(2):356-363. doi: 10.1177/1932296817731422. Epub 2017 Sep 26. PMID 28946756
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com